CLINICAL TRIAL: NCT01331889
Title: Potassium Change in the Fluid Management System (FMS) Reservoir and Its Effect on the Plasma Potassium Concentration During Liver Transplantation Surgery
Brief Title: Effect of Rapid Transfusion With Fluid Management System (FMS) on Plasma Potassium in Liver Transplantation Recipients
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Collaborators: Seoul National University (Other)
Responsible Party: Principal Investigator, Chul-Woo Jung, Assistant Professor, Seoul National University Hospital
Other Study IDs: FMS_potassium
Record Dates: First submitted 2011-04-05; First posted 2011-04-08 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Condition Requiring Rapid Transfusion During Liver Transplantation Surgery
Keywords: transfusion; liver transplantation; potassium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Potassium concentration: plasma potassium concentrations in the Fluid Management System (FMS) reservoir, arterial blood, and central venous blood

SUMMARY:
Rapid infusion of red blood cells is known to result in hyperkalemia in the body. However, potassium concentration in the blood mixture (usually made of RBC, FFP and normal saline) in the reservoir of rapid infusion system and its effect on the plasma potassium change during rapid transfusion are unknown. This study is designed to investigate these changes while massive transfusion is performed during liver transplantation surgery.

ELIGIBILITY:
Inclusion Criteria:

* preoperative anemia (hemoglobin < 10 g/dl)
* preoperative coagulopathy

Exclusion Criteria:

* children under age 18
* low risk of intraoperative bleeding

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult liver transplantation recipients
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2011-10; Primary Completion 2015-03 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
potassium concentration in the Fluid Management System (FMS) reservoir | after transfusion of 150 ml of blood mixture
  During bolus transfusion (300ml) of blood mixture, blood sample is taken from the side port of infusion line of Fluid Management System (FMS) when 150 ml of blood mixture was transfused. Because the priming volume of the internal circuit is approximately 100 ml, blood sample that was taken after 150 ml transfusion represents the content in the reservoir.

SECONDARY OUTCOMES:
plasma potassium of the patient | before and after transfuison of 300 ml of blood mixture
  Just before transfusion starts, blood samples are taken from the central venous catheter and arterial line at the same time to measure baseline values. At the immediate end of transfusion, blood samples are taken again from the same sites to measure the resultant changes.

CONTACTS AND LOCATIONS:
Overall Officials: Chul-Woo Jung, MD. PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea